CLINICAL TRIAL: NCT03587831
Title: Vertical Sleeve Gastrectomy and Lifestyle Modification for the Treatment of Non-Alcoholic Steatohepatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURG-2018-26636
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VSG + LSM (Experimental): Procedure/Surgery: Vertical Sleeve Gastrectomy will be performed using five laparoscopic ports. The short gastric and epiploic vessels will be taken down With a 40 French Bougie in place, the greater curvature will be excised starting 6 cm proximal to the pylorus.
  Behavioral: Lifestyle Modification Counseling - The intensive lifestyle intervention will align with methods listed in the LSM arm description. However, participants assigned to the VSG will not have calorie ceilings during the first 6 months of rapid weight loss, and they will receive additional instruction regarding food volume and adequate protein intake.
  Interventions: Procedure: Vertical Sleeve Gastrectomy; Behavioral: Lifestyle Modification Counseling
- LSM (Active Comparator): Behavioral: Lifestyle Modification Counseling - The intensive lifestyle intervention is modeled after the LookAHEAD trial, with modules modified for participants undergoing surgery, and designed to produce maximum achievable weight loss. Both groups will increase their level of moderate-intensity physical activity (such as walking) to a total of 325 minutes per week. All lifestyle-medical management participants will be given calorie intake targets of 1200, 1500, or 1800 kilocalories per day, depending on body weight, with the goal of producing a weight loss of 1 to 2 pounds per week. There will be 24 weekly counseling meetings during the first 6 months, bi-weekly meetings between months 7 and 9, and monthly meetings between months 10 and 12.
  Interventions: Behavioral: Lifestyle Modification Counseling

INTERVENTIONS:
Procedure: Vertical Sleeve Gastrectomy — Surgical Procedure: Vertical Sleeve Gastrectomy
  Arms: VSG + LSM
Behavioral: Lifestyle Modification Counseling — Behavioral Intervention: Lifestyle Modification Counseling

SUMMARY:
Participants meeting study entry criteria are randomized with equal probability to one of two study groups: (1) Lifestyle modification or (2) Vertical Sleeve Gastrectomy (VSG) with Iifestyle modification, followed for 12 months. The primary goal for the trial is to determine if the investigators can recruit, randomize, and retain participants to perform invasive and non-invasive measurements of NASH and fibrosis, deliver lifestyle modification and demonstrate the safety of VSG. The investigators wish to also understand which of these two interventions is more effective in achieving, 12 months after entry into the trial, a reduction in NAS composed of the non-weighted scores: (1) steatosis 0-3 (2) Inflammation 0-3 and (3) ballooning 0-2. Secondary goals include comparing the two treatment groups for changes in other measured outcomes including MRI assessments of intrahepatic triglyceride and liver elasticity and serum markers. As a pilot study, a sample size of 20 in each group should offer significant information as to the difference in NAS score reduction between to two groups and achieve adequate power to distinguish clinically significant changes in the primary and secondary outcome measures. These data support the overarching objective i.e. to provide evidence that a larger, longer-term clinical outcomes trial is feasible. A goal is for a longer term follow up for 5 years to assess the durability of treatment effects and treatment differences.

DETAILED DESCRIPTION:
The pilot study proposed in this protocol will determine whether patients with a BMI of 35-60 kg/m2 will consent to liver biopsy, accept randomization to VSG, participate in lifestyle modification for a one-year period and consent to a paired liver biopsy at 12 months. Candidates will be biopsied with 48 randomizations within the first year yielding 20 (including dropouts) participants/group. This should be sufficient to further estimate meaningful differences in liver histology given the estimated weight loss of lifestyle modification with and without VSG and a correlation of percent weight loss and histological score improvement over the short term (12 months). Determining the impact of the VSG is essential for expanding the traditional indications for bariatric surgery and thus, broadening the potential impact of this pilot study.

The investigators will screen patients by telephone between the ages of 30 and 70 with a self-reported BMI of 35-60 kg/m2, a history of prediabetes, or type 2 diabetes. Prospective participants will be asked to provide a copy of their most recent liver chemistries to see if the AST or ALT fall in the inclusion range. The investigators will screen for a history of alcohol or other substance abuse and a surgical history that would preclude a safe VSG. Prospective participants will be invited to attend a seminar. They will be instructed to keep a food and exercise log for two weeks and return for a second visit. After consent is signed, during the eligibility review period participants will have their height and weight recorded, history reviewed, liver function tests, HbA1c, a urine sample, a basic metabolic profile, and INR will be obtained at this time and the participant will be referred for a liver biopsy. If the biopsy is consistent with NASH with a NAS >=4, then the participant will undergo MRI assessment and serum markers for inflammation. Vital signs (pulse, temperature, respiration, blood pressure, weight and BMI) will be obtained at each study visit. Participants will then begin an 800 calorie per day diet for 7 days during which they will receive their randomization assignment to VSG or not; all participants will receive lifestyle modification as the investigators need to see if surgery can provide any additional benefit to lifestyle modification. A basic metabolic panel will be performed at the conclusion of the 800 calorie diet. VSG will be performed laparoscopically and the greater curvature resected 6 cm for the pylorus to the angle of His over a 40 French Bougie. Lifestyle modification can begin immediately after surgery, though the VSG participants will not have calorie limits until 6 months after surgery. Participants will be seen regularly by the hepatologist and surgeon at 1 week, 4 weeks, 12 weeks, 6 months, and 12 months. Lifestyle will be delivered on an individual basis once per week for the first 6 months, twice per month for the next 3 months, and monthly up to one year. Vitamins A, B1, B12 and D and a comprehensive metabolic panel including liver chemistries will be performed at 3 months and 12 months in both groups. At 12 months a repeat liver biopsy will be performed (participants will have the opportunity to select an alternative approach if they did not have a good experience with the initial liver biopsy in order to ensure a paired specimen). This decision will be made in conjunction with the interventional radiologist. MRI for steatosis and elasticity will be performed and serum inflammatory and fibrosis markers will be obtained at 12 months as well as the collection of another urine sample. Participants will exit the study but will continue usual care after 12 months. We will create a biorepository for stool samples to measure the microbiome and for remaining liver tissue to measure the transcriptome.

Participants meeting study entry criteria are randomized with equal probability to one of two study groups: (1) Lifestyle modification (LSM) or (2) Vertical Sleeve Gastrectomy (VSG + LSM) with Iifestyle modification, followed for 12 months. The primary goal for the trial is to determine if we can recruit, randomize, and retain participants to perform invasive and non-invasive measurements of NASH and fibrosis, deliver lifestyle modification and demonstrate the safety of VSG. The investigators wish to also understand which of these two interventions is more effective in achieving, 12 months after entry into the trial, a reduction in NAS composed of the non-weighted scores: (1) steatosis 0-3 (2) Inflammation 0-3 and (3) ballooning 0-2. Secondary goals include comparing the two treatment groups for changes in other measured outcomes including MRI assessments of intrahepatic triglyceride and liver elasticity and serum markers. As a pilot study, a sample size of 20 in each group should offer significant information as to the difference in NAS score reduction between to two groups and achieve adequate power to distinguish clinically significant changes in the primary and secondary outcome measures. These data support the overarching objective i.e. to provide evidence that a larger, longer-term clinical outcomes trial is feasible. A goal is for a longer term follow up for 5 years to assess the durability of treatment effects and treatment differences.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 70 years at eligibility visit.
* At least one of the following:
* Diagnosed with NASH with a total NAS ≥ 4 including a ballooning score of at least 1
* Diagnosed with T2DM or prediabetes, HbA1c< 9%
* Body Mass Index (BMI): 35.0-60.0 kg/m2 at eligibility visit.
* Willingness to accept random assignment to either treatment group.
* All patients must have insurance with no exclusion for obesity related treatments or management of obesity surgery complications. This applies to all participants enrolled in the study
* Evidence of liver fat present in the baseline MR images
* Suitable for liver biopsy
* Willingness to comply with the follow-up protocol and successful completion of the run-in (described below).
* Written informed consent.
* English speaking

Exclusion Criteria:

* Cardiovascular event (myocardial infarction, acute coronary syndrome, coronary artery angioplasty or bypass, stroke) in the past six months.
* Current evidence of congestive heart failure, angina pectoris, or symptomatic peripheral vascular disease.
* Pulmonary embolus or thrombophlebitis in the past six months.
* Cancer of any kind (except basal cell skin cancer or cancer in situ) unless documented to be disease-free for five years.
* Significant anemia (hemoglobin 2.0 g/dL or more below normal range) or history of coagulopathy. (Low range for women would be 10, low range for men would be 11)
* Serum creatinine >1.8 mg/dL.
* Serum total bilirubin greater than the upper limit of normal in the absence of Gilbert's syndrome, or alkaline phosphatase or ALT or AST greater than 2.5x the upper limit of normal. Elevated INR.
* Alcohol intake more than one drink or >20 grams per day
* History of stomach surgery, bile duct surgery, pancreatic surgery, splenectomy, or colon resection.
* Gastric or duodenal ulcer in the past six months.
* History of intra-abdominal sepsis (except for uncomplicated appendicitis or diverticulitis more than six months prior to enrollment).
* Previous organ transplantation.
* Self-reported HIV-positive status, active tuberculosis, active malaria, chronic hepatitis B or C, cirrhosis, or inflammatory bowel disease.
* Currently pregnant or nursing, or planning to become pregnant in the next two years.
* History of alcohol, drug, or opioid dependency (excluding nicotine) in the past five years.
* Active psychosocial or psychiatric problem that is likely to interfere with adherence to the protocol.
* A score of 17 or greater on the CES-D questionnaire administered on a typical week for the participant.
* Presence of any chronic or debilitating disease that would make adherence to the protocol difficult.
* Serum c-peptide <1.0 ng/ml post prandial.
* Exclusions may also be made at the discretion of the attending physician or the eligibility committee.
* History of endoscopy demonstrating esophagitis or Barrett's changes in the esophagus.
* Any history of dysphagia.
* Fibrosis score > 3
* Use of Rezdiffra (resmetirom).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Histologic improvements in NAFLD Activity Score (NAS) | Month 12
  The scale used is NAS - this is the NAFLD (Nonalcoholic Fatty Liver Disease) Activity Score.
  The NAS was developed to provide a numerical score for patients who most likely have NASH. Accordingly, NAS is the sum of the separate scores for steatosis (0-3), hepatocellular ballooning (0-2) and lobular inflammation (0-3). NAS scores of 0-2 are largely considered not diagnostic of NASH, scores of 3-4 are often considered not diagnostic, borderline, or potentially positive for NASH. Scores of 5-8 are largely considered diagnostic of NASH.
  It is expected that the addition of VSG to lifestyle modification will result in more robust histologic improvements in NAFLD Activity Score (NAS) compared to lifestyle modification alone.

CONTACTS AND LOCATIONS:
Overall Officials: Sayeed Ikramuddin, M.D., M.H.A., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of San Fransisco, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota